CLINICAL TRIAL: NCT05966922
Title: Effects of Transcutaneous Electrical Stimulation on the Sinoatrial Node Function
Brief Title: Transcutaneous Electrical Stimulation & Sinoatrial Node Function
Acronym: TENS&HR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ISTPMRTENS1
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Electricity; Effects; Heart Arrhythmia
Keywords: Transcutaneous electrical nerve stimulation; Neuromuscular electrical stimulation; Heart rhythm; heart rate variability
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This study will be conducted in an experimental study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrical Stimulation (Experimental): Electrical Stimulation and Sham will be delivered transcutaneously in random consecutive sessions
  Interventions: Procedure: Transcutaneous Electrical Stimulation

INTERVENTIONS:
Procedure: Transcutaneous Electrical Stimulation — Electrical Stimulation and a sham will be administered through the skin in random consecutive sessions in a study group. A single monophasic square electrical pulse and transcutaneous electrical nerve stimulation will be applied to the forearm volar aspect.

SUMMARY:
Transcutaneous electrical stimulation (TES) is used in clinical practice to diagnose or treat a diverse range of medical conditions for over a century. Although the benefits of TES are well known, its potential side effects on the heart have not been convincingly clarified. This study will test whether TES has any effect on the sinoatrial node (SAN).

DETAILED DESCRIPTION:
It was hypothesized that: 1) TES has effects indirectly via peripheral afferents or directly on the SAN, and 2) TES causes a change in the R-R interval (HRV). The aim of this study was to test these hypotheses.

This research protocol will have three phases: first, the effect of a single electrical pulse on heart rate variability (HRV) will be examined in Experiment I. The effects of conventional TENS and acupuncture-like TENS on HRV will be also investigated in Experiment II. Finally, the effect of time and rest on the HRV will be tested in Experiment III. Subjects will be in a sitting position with 90-degree flexion at the elbow and supination of the hand during electrical stimulation. A pair of square (4 x 4 cm), self-adhesive, pre-gelled skin electrodes will be used for stimulation. The electrodes will be placed over the flexor aspect of the right forearm. Three-lead electrocardiogram (ECG) recording will be obtained to determine the change of HRV during rest and electrical stimulation sessions. The participant's ECG data will be continuously captured by noninvasive sensors [self-adhesive pre-gelled Ag/AgCl surface electromyography (sEMG) electrodes, Redline® Istanbul, Türkiye] transmitted through a data acquisition system.

The main outcome variable is the heart rhythm. In this context, electrical stimulus-related QRS wave and RR interval change (heart rate variability) will be examined. The possible direct effect of an electrical stimulus on the appearance of the QRS wave will be investigated in the time domain using the Peristimulus time histogram and the Waveform average technique. ECG data will be analyzed using a software package (Cambridge Electronic Designs, Cambridge, UK).

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adult volunteer

Exclusion Criteria:

* Pregnancy
* Alcohol or drug abuse,
* Any medication with potential effects on the cardiovascular system

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | up to 2 weeks
  RR interval will be calculated
Heart rate variability | up to 2 weeks
  Variability of RR interval will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: İLHAN KARACAN, MD, Prof, Study Chair — İstanbul Physical Therapy Rehabilitation Training & Research Hosptial
Locations (1):
- İstanbul Physical Therapy Training and Research Hospital, Istanbul, Turkey (Türkiye)